CLINICAL TRIAL: NCT05687851
Title: A Single-arm, Multicenter, Phase II Study to Evaluate Cadonilimab（AK104） Combined With Radiotherapy For The Treatment of Locally Advanced Cervical Cancer
Brief Title: Study Of Cadonilimab Combined With Radiotherapy In The Treatment of Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); Henan Cancer Hospital (Other Government); Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qi Zhou, Professor, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG010
Record Dates: First submitted 2022-12-24; First posted 2023-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: Local advanced cervical cancer; Concurrent chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Participants receive Cadonilimab at a dose of 10 mg/kg, Q3W (Day 1 of each 21 day treatment cycle) via IV infusion, until disease progression, intolerable toxicity, investigator determines that the participant cannot continue to benefit, withdraw informed consent, or Cadonilimab treatment over 2 years. During the q3w dosing period of Cadonilimab, participants receive radiotherapy including external beam radiotherapy (EBRT) and followed by brachytherapy.
  Interventions: Drug: Cadonilimab（AK104）; Radiation: EBRT; Radiation: BT

INTERVENTIONS:
Drug: Cadonilimab（AK104） — q3w iv
Radiation: EBRT — 45-50.4Gy
Radiation: BT — ≥80Gy

SUMMARY:
Cadonilimab（AK104）is a humanized IgG1 bispecific antibody that targets PD-1 and CTLA-4.

This is a single-arm, multicenter, open-label, phase II study, the purpose of this study is to evaluate the efficacy and safety of Cadonilimab plus radiotherapy in participants with locally advanced cervical cancer who do not tolerate chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign written informed consent.
2. Women aged ≥18 years at the time of study entry.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0-2.
4. Life expectancy ≥12 weeks.
5. Intolerance to chemotherapy regimens.
6. Histologically confirmed cervical cancer.

   1. Histologically-confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix;
   2. Not receiving systemic anti-tumour therapy (including but not limited to radiotherapy, targeted therapy and immunotherapy, etc; concurrent chemotherapy is not included. Note: Removal or biopsy of pelvic lymph nodes or para-aortic lymph nodes for the purpose of clinical staging is allowed).
   3. Locally advanced cervical cancer（LACC）: The International Federation of Gynecology and Obstetrics (FIGO) 2018 Stage IB3/IIA2, IIB-IVA.
7. At least one measurable tumor lesion according to RECIST v1.1 criteria.
8. Available archived tumor tissue samples or recent biopsies.
9. Adequate organ function.
10. For fertile women with negative serum pregnancy and effective contraception within 7 days before administration (until 120 days after the last administration of the study drug and at least 180 days after radiotherapy)

Exclusion Criteria:

1. Other histological types of cervical cancer (eg, neuroendocrine carcinoma, small cell carcinoma, sarcoma, etc).
2. Evidence of distant metastases.
3. Have received total hysterectomy.
4. Subject with other active malignancies within 2 years prior enter the study.
5. Subject who cannot receive brachytherapy.
6. Active or prior documented autoimmune disease that may relapse.
7. History of interstitial lung disease or noninfectious pneumonitis.
8. Subject with the clinically significant cardio-cerebrovascular disease.
9. History of severe hypersensitivity reactions to other mAbs.
10. Prior allogeneic stem cell transplantation or organ transplantation.
11. Subjects who require systemic treatment with glucocorticoid (>10 mg/day of prednisone or equivalent glucocorticoid) or other immunosuppressive agents within 14 days prior enter the study.
12. Receipt of live attenuated vaccines within 30 days prior to the first dose of the study drug.
13. Prior exposure to any experimental antitumor vaccines, or any agent targeting T-cell costimulation or immune checkpoint pathways (eg, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, anti-CD137 or anti-OX40 antibody, etc).
14. Any condition that, in the opinion of the Investigator, would interfere with the evaluation of the study drug or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by Investigator | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR per RECIST v1.1.

SECONDARY OUTCOMES:
DCR | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
PFS | Up to approximately 30 months
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
OS | Up to approximately 40 months
  OS is the time from randomization to death due to any cause
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status Score and Physical Function Score. | Baseline and up to approximately 40 months
  The EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Global scores are converted to a score of 0 to 100, with a higher score indicating improved health status. The change from baseline in EORTC QLQ-C30 score will be presented.
Number of participants with adverse events (AEs) | Up to approximately 40 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhou, MD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing university Cancer Hospital, Chongqing, CHN, China

IPD SHARING:
Plan to Share IPD: No